CLINICAL TRIAL: NCT06128122
Title: Dextrose Concentration Decline Rate in Vivo After Intraarticular Knee and Subcutaneous Injection
Brief Title: Dextrose Concentration Decline Rate in Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Dean Reeves Clinic (Other)
Responsible Party: Principal Investigator, Dr. Dean Reeves, Principal Investigator, Dr. Dean Reeves Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Reeves-DexConc01
Record Dates: First submitted 2023-11-01; First posted 2023-11-13 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Dextrose Concentration
Keywords: Dextrose; Hydrodissection; Proliferation
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Dextrose curve production from a single individual
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dextrose injection intraarticularly and in subcutaneous tissue with timed dextrose measurements (Experimental): Step One: Injection of 30 ml of D12.5% in the knee anteromedially with knee flexed. Placement of IV catheter into the suprapatellar pouch, and secure catheter. Withdraw and analyze samples for dextrose levels at 15-minute intervals. If catheter fails, aspirate directly from suprapatellar pouch.
  Step Two: Inject 1-3 ml of D5W into interstitial space about a functioning Dexcom G7 sensor. Measure dextrose levels every 5 minutes on a Dexcom receiver.
  Interventions: Procedure: Intrarticular and subcutaneous dextrose injection with timed measurement of dextrose levels

INTERVENTIONS:
Procedure: Intrarticular and subcutaneous dextrose injection with timed measurement of dextrose levels — Step one: 30 mL of 12.5%/0.1% lidocaine will be injected into the knee using an inferomedial approach. Using ultrasound guidance, a 20-gauge 2-inch I.V. catheter will be placed in the suprapatellar pouch, by which samples of synovial fluid from the pouch will be withdrawn and analyzed for glucose level.
  Step two: 3 mL of D5W will be injected into a marked spot on the back of the upper arm. A sensor/transmitter (Dexcom G7 Dexcom) is placed at the site of injection. The sensor/transmitter will begin providing dextrose levels at 5 minute intervals beginning one-half hour after placement of the sensor/transmitter, transmitted to a paired smart phone.
  Other Names: Glucose injection (Dextrose is the form of glucose that humans can metabolize)

SUMMARY:
Measuring the speed of decrease in dextrose concentration to help design more accurate in vitro studies

DETAILED DESCRIPTION:
Rationale: In vitro studies of the potential mechanism of action of therapeutic dextrose injection commonly place human or animal cells in a dextrose (glucose) culture medium for a prolonged period of time, typically 24 hours, and expose them to high dextrose levels, typically 1-25% (1000- 25,000mg%). High glucose levels in culture media can cause cell death. Given that cellular apoptosis/death has not been shown to occur after therapeutic dextrose injection in vivo by histologic analysis, we expect that elevated glucose levels drop rapidly in vivo. In this study 12.5% dextrose will be injected intraarticularly (in the knee) and dextrose 5% will be injected subcutaneously, and dextrose level measurements will be obtained at timed intervals after each in order to produce a curve depicting the pattern and speed of decrease in dextrose levels after in vivo injection. In vitro studies can then utilize this information to alter the pattern and speed of decrease of dextrose levels to mimic in vivo conditions, and in so doing provide more useful data on potential mechanisms of therapeutic dextrose injection in soft tissue and joints.

ELIGIBILITY:
Inclusion Criteria:

Able to be relatively immobile for intermittent measurement of dextrose levels

Exclusion Criteria:

Diabetic

Ages: 69 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Dextrose levels in synovial fluid | 0.5, 1, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, and 6.0 hours
  Dextrose level in synovial fluid of the knee, beginning 1/2 hour after intraarticular injection
Dextrose level in subcutaneous tissue (interstitial space) in upper arm or abdomen | Continuous glucose measurement
  Dextrose levels at time zero and every 5 minutes after injection subcutaneously

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Reeves, M.D., Principal Investigator — Dr. Dean Reeves Clinic
Locations (1):
- Kenneth Dean Reeves, Shawnee Mission, Kansas, United States

IPD SHARING:
Plan to Share IPD: No